CLINICAL TRIAL: NCT04846192
Title: Prognosis of Nutritional Status for Surgical Peri Hilar Cholangiocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PI058
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Perihilar Cholangiocarcinoma
Keywords: sarcopenia; nutritional status; surgery
MeSH Terms: conditions — Klatskin Tumor; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Other: Nutritional evaluation

INTERVENTIONS:
Other: Nutritional evaluation — Collecting existing data on pre operative nutritional status and outcomes after surgery

SUMMARY:
Curative treatment of peri hilar cholangiocarcinomas is R0 surgery and require major hepatectomy with biliary tract resection. These complexe procedures can lead to high morbidity and mortality. A severe alteration of nutritional status before the surgery might be a poor prognosis for survival.

DETAILED DESCRIPTION:
Peri hilar cholangiocarcinomas are rare tumors, which when diagnosed at the resectable stage, require major hepatic resection associated with biliary reconstruction. These are complex procedures with a high morbidity and mortality, mainly due to postoperative hepatic failure and sepsis.

These patients undergo optimization of liver function with portal embolization according to the volume of the future remaining liver and preoperative biliary drainage. On top of technical challenges of the surgery, the patients usually present a significant alteration of the general condition at the time of diagnosis, with denutrition that can be severe. The importance of evaluating the preoperative nutritional status in the context of oncological surgery is increasingly recognized in the literature. Different nutritional scores exist such as the CONUT score, PNI, or the evaluation of sarcopenia on imaging examinations and have shown an impact on morbi-mortality in liver surgery.

ELIGIBILITY:
Inclusion Criteria:

* Surgical peri hilar cholangiocarcinoma from 01/01/2003 to 04/01/2021 at Nancy University Hospital

Exclusion Criteria:

* Non curative surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical peri hilar cholangiocarcinoma at Nancy University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 01/01/2003 to 04/01/2021
Disease Free Survival | 01/01/2003 to 04/01/2021

SECONDARY OUTCOMES:
Morbidity | 01/01/2003 to 04/01/2021
  Post operative complications : Dindo-Clavien > or = 3

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Ayav, PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Otsuji H, Yokoyama Y, Ebata T, Igami T, Sugawara G, Mizuno T, Nagino M. Preoperative sarcopenia negatively impacts postoperative outcomes following major hepatectomy with extrahepatic bile duct resection. World J Surg. 2015 Jun;39(6):1494-500. doi: 10.1007/s00268-015-2988-6. PMID 25651963
- [Background] Golse N, Nunez J, Mazzotta A, Cano L, Bergeat D, Sulpice L, Jeddou H, Abdelrafee A, Sa Cunha A, Cherqui D, Adam R, Boudjema K, Vibert E. Personalized Preoperative Nomograms Predicting Postoperative Risks after Resection of Perihilar Cholangiocarcinoma. World J Surg. 2020 Oct;44(10):3449-3460. doi: 10.1007/s00268-020-05618-8. PMID 32474628
- [Background] Cruz-Jentoft AJ, Sayer AA. Sarcopenia. Lancet. 2019 Jun 29;393(10191):2636-2646. doi: 10.1016/S0140-6736(19)31138-9. Epub 2019 Jun 3. PMID 31171417
- [Result] Yugawa K, Itoh S, Kurihara T, Yoshiya S, Mano Y, Takeishi K, Harada N, Ikegami T, Soejima Y, Mori M, Yoshizumi T. Skeletal muscle mass predicts the prognosis of patients with intrahepatic cholangiocarcinoma. Am J Surg. 2019 Nov;218(5):952-958. doi: 10.1016/j.amjsurg.2019.03.010. Epub 2019 Mar 14. PMID 30902342